CLINICAL TRIAL: NCT04861961
Title: Prospective Randomized Study Comparing Three Hypoabsortive Techniques for the Treatment of Type IV Obesity: Double-anastomosis Duodenal Switch (DS), Single- Anastomosis Duodenal Switch SADI-S) and One Anastomosis Gastric By-pass (OAGBP)
Brief Title: Comparison of Three Hypoabsortive Surgical Techniques for Treatment of Type IV Morbid Obesity
Acronym: BAR-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Javier Osorio, Dr. Javier Osorio, MD, PhD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAR-3
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Bariatric Surgery; Morbid Obesity
Keywords: Bariatric Surgery; Morbid Obesity; Hypoabsortive surgery; Duodenal Switch; SADI-S; One-anastomosis gastric by-pass; Gastro-esophageal reflux
MeSH Terms: conditions — Obesity, Morbid; Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Prospective randomized study comparing three bariatric surgical techniques
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laparoscopic duodenal switch (DS) (Active Comparator): Standard duodenal switch (double anastomoses). Roux-en-Y reconstruction.
  Interventions: Procedure: DS vs. SADI-S vs. OAGBP
- Laparoscopic Single Anastomosis Duodenum-Ileal bypass with Sleeve gastrectomy (SADI-S) (Active Comparator): Simplified duodenal switch with one anastomosis. Duodeno-ileal omega reconstruction ("Billroth II-like").
  Interventions: Procedure: DS vs. SADI-S vs. OAGBP
- Laparoscopic one anastomosis gastric bypass (OAGBP) (Active Comparator): Gastric bypass of one anastomoses. Gastro-jejunal omega reconstruction (Billroth II).
  Interventions: Procedure: DS vs. SADI-S vs. OAGBP

INTERVENTIONS:
Procedure: DS vs. SADI-S vs. OAGBP — Randomizacion of candidates for either conventional DS, SADI-S or OAGBP.

SUMMARY:
Morbid obesity is the first non-traumatic cause of death in the western population and it is also progressively beginning to affect the developing countries. Bariatric surgery provides better results than pharmacological treatments and lifestyle changes, granting a better control of comorbidities.

Duodenal switch (DS) has proben to be the most effective surgical treatment for grade IV morbid obesity and its comorbidities. However, it is not widely used due to its technical complexity and the risk of long-term complications. Single Anastomosis Duodenum-Ileal bypass with Sleeve gastrectomy (SADI-S) was concieved in 2007 as a one-anastomosis simplification of DS, intended to diminish the surgical time and postoperative risks. Recently, another simplified hypo-absorptive technique has started to be widely used: the one anastomosis gastric bypass (OAGBP), also called mini-gastric gypass. It consists of a gastric pouch associated with a gastro-jejunal anastomosis in omega (Billroth II). Despite the potential advantages of these emerging surgical techniques (SADI-S and OAGBP), there is no solid evidence on its efficacy for the treatment of grade IV obesity in comparison with DS. Besides, there is also there is a lack of studies reporting on prospective acid and bile reflux after omega digestive reconstructions, suche as "Billroth II-like" (SADI-S) and "Billroth II" (OAGBP). Bile reflux is potentially premalignant condition.

This prospective randomized study aims to compare conventional DS with SADI-S and OAGBP. We include all morbidly obese patients with BMI ≥ 50 kg/m2 aged 18 years or more. Exclusion criteria are patients who do not fulfill our preoperative bariatric assessment for surgery and those with contraindications for hypo absorptive or mixed surgery.

The main objective of the study is to compare the percentage of excess weight lost at 2 and 5 years after the three different surgical procedures. As a secondary objective, gastroesophageal reflux (GERD) will be compared before and 2 years after surgery, based on GERD symptoms test, gastroscopy and a esophageal pH-impedanciometry in selected patients. Other secondary objectives are comparison of short-term complications, metabolic comorbidities, depositional habit, quality of life and metabolic and nutritional deficiencies at two years of surgery.

DETAILED DESCRIPTION:
Morbid obesity is the first non-traumatic cause of death in the western population and it is also progressively beginning to affect the developing countries. Bariatric surgery provides better results than pharmacological treatments and lifestyle changes, granting a better control of comorbidities.

Duodenal switch (DS) has shown to be the most effective surgical treatment for morbid obesity and its comorbidities. However, it is not widely used due to its technical complexity and the risk of long-term complications. In 2007 Drs. Sánchez-Pernaute and Torres introduced a simplified version of the DS technique: Single Anastomosis Duodenum-Ileal bypass with Sleeve gastrectomy (SADI-S). SADI-S consists of a vertical gastrectomy (VG) and a duodenum-ileal anastomosis preserving the pylorus with jejunal exclusion and a total common-alimentary loop originally of 200 cm and later standardized to 300 cm to reduce the risk of nutritional deficits. In order to diminish the surgical time and postoperative risks an omega reconstruction is performed without an ileo-ileal anastomosis. SADI-S can be performed either directly as primary surgery, planned in two stages, or as revisional surgery in case of insufficient weight loss or weight regain after VG. In terms of weight loss and comorbidity resolution, SADI-S' reported results are similar to those reported in historical DS series, but no prospective comparative studies have been published.

Recently, another simplified hypo-absorptive technique has started to be widely used: the one anastomosis gastric bypass (OAGBP), also called mini-gastric gypass. It consists of a gastric pouch associated with a gastro-jejunal anastomosis (Billroth II). It was initially described by R. Rutledge in 1997 and despite its first publication was in 2001, only lately it has been approved as a standard bariatric technique. OAGBP with a 200 cm biliopancreatic limb has shown good results in weight loss and control of comorbidities, higher than those achieved by VG and proximal Roux-en-Y gastric bypass (RYGBP) with 50 cm biliopancreatic limb and 150 cm alimentary limb, as it has been demonstrated in two prospective randomized studies and a recent meta-analysis. However, the OAGB results have not been compared with other hypo absorptive surgical techniques, such as DS or SADI-S.

In comparison to the DS, which has a Y-Roux reconstruction, SADI-s and OAGBP have a "Billroth II-like" or omega reconstruction. Despite the potential advantages of these emerging surgical techniques, bile reflux is the main issue of omega reconstructions. In our most recently published series including 440 consecutive patients, we reported that 1.7% of patients required conversion to DS due to symptomatic bile reflux. It would be reasonable to expect higher incidence of bile reflux in techniques with omega reconstruction that do not preserve the pyloric barrier, such as OAGBP. However, some authors claim that with a 200 cm biliopancreatic limb most of the bile is reabsorbed by the intestine before it reaches the gastro-jejunal anastomosis. This would minimize bile reflux in comparison to the historical series of Billroth II reconstruction after gastrectomy for oncological or peptic disease (in which the biliopancreatic loop is much shorter, generally around 50 cm). Reported incidences of symptomatic bile reflux after OAGBP vary between 0.5% and 1.5%, comparable to our SAID-S results. It is worth mentioning that not all bile refluxes are symptomatic and that biliary gastritis is a premalignant condition. At present, there is a lack of literature on acid and bile reflux after bariatric surgery comparing the 3 digestive reconstruction techniques: (i) Roux-en-Y with pyloric preservation (DS), (ii) omega reconstruction with pyloric preservation or "Billroth II-like" (SADI-S) and (iii) omega reconstruction without pyloric preservations or Billroth II (OAGBP).

This prospective randomized study aims to compare conventional DS with SADI-S and OAGBP. We include all morbidly obese patients with BMI ≥ 50 kg/m2 and candidates to a directly DS following our treatment algorithm. Exclusion criteria are patients who do not fulfill our preoperative bariatric assessment for surgery and those with contraindications for hypo absorptive or mixed surgery.

The main objective of the investigation is to compare the percentage of excess weight lost at 2 and 5 years after the three different surgical procedures. For the study of weight evolution, both Dietetics' and General Surgery's postoperative standardized routine controls at our outpatient centre will be used.

As a secondary objective, gastroesophageal reflux (GER) will be compared before and 2 years after surgery. A GER's symptoms test, gastroscopy and a esophageal pH-impedance analysis in selected patients will be employed. Other secondary objectives include the comparison of short-term complications, metabolic comorbidities, bowel habit and quality of life two years after the surgical procedure. Furthermore, a medium and long term follow up on metabolic and nutritional deficiency will be performed.

For the morbidity and mortality analysis, the patients' electronic medical history records will be revised. Short postoperative complications (up to 30th postoperative day) will be classified according to Clavien-Dindo classification. Comorbidities' evolution will be evaluated following our centre follow-up protocol before and annually after the surgery. Data will be collected in a prospective database. The quality-of-life study will be carried out with the SF-12 test. The metabolic and nutritional deficit analysis will be carried out through the annual analytical data collected during the follow-up of the patients according to common clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 and younger than 65 who fulfil bariatric surgery indications
* BMI between 50 and 60 kg / m2
* Patients with a good overall condition to perform a one step surgery
* Signing up of the informed consent for the study
* Patient suitable for laparoscopic surgery

Exclusion Criteria:

* Previous bariatric surgery
* Two stage surgery
* Medical contraindication for a hypoabsorptive surgery due to previous pathology: inflammatory bowel disease, organ transplantation or candidate for a transplant, previous intestinal resection surgery
* Conversion to laparotomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Percentage of excess weight lost (% EWL) | At 5 years after surgery
  % EWL considering ideal BMI = 25 kg/m2

SECONDARY OUTCOMES:
Gastroesophageal reflux | 2 years after surgery
  Gastroesophageal reflux as defined by the Lyon Consensus
Postoperative complications | 30 days after surgery
  Complications will be recorded according to the Clavien-Dindo classification
Postoperative mortality | 90 days after surgery
  Short-term mortality after surgery
Metabolic comorbidities | At 5 years of surgery
  Comorbidities related to metabolic syndrome and morbid obesity: Type-2 diabetes (DM2), arterial hypertension (HT), dyslipidemia (DLP) and obstructive sleep apnea (OSA).
Quality of life (SF-12 test) | At 2 years of surgery
  Quality of life determined by the SF-12 test
Depositional habit | At 2 years of surgery
  The number of depositions per day, the consistency of the depositions according to the Bristol visual scale and faecal incontinence and / or defecation urgency according to Wexner Vaixey scale
Need of revisional surgery | At 5 years of surgery
  Revisonal surgery due to nutritional defficiencie, gastroesophageal reflux or other causes

CONTACTS AND LOCATIONS:
Overall Officials: Javier Osorio, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitary de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
On demand to IP
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: April 2026 to april 2027
Access Criteria: On demand to PI

REFERENCES:
- [Background] Finno P, Osorio J, Garcia-Ruiz-de-Gordejuela A, Casajoana A, Sorribas M, Admella V, Serrano M, Marchesini JB, Ramos AC, Pujol-Gebelli J. Single Versus Double-Anastomosis Duodenal Switch: Single-Site Comparative Cohort Study in 440 Consecutive Patients. Obes Surg. 2020 Sep;30(9):3309-3316. doi: 10.1007/s11695-020-04566-5. PMID 32240495
- [Background] Sorribas M, Casajoana A, Sobrino L, Admella V, Osorio J, Pujol-Gebelli J. Experience in biliopancreatic diversion with duodenal switch: results at 2, 5 and 10 years. Cir Esp (Engl Ed). 2021 Feb 13:S0009-739X(21)00030-0. doi: 10.1016/j.ciresp.2021.01.008. Online ahead of print. English, Spanish. PMID 33593597
- [Background] Admella V, Osorio J, Sorribas M, Sobrino L, Casajoana A, Pujol-Gebelli J. Direct and two-step single anastomosis duodenal switch (SADI-S): Unicentric comparative analysis of 232 cases. Cir Esp (Engl Ed). 2021 Aug-Sep;99(7):514-520. doi: 10.1016/j.cireng.2021.06.017. Epub 2021 Jul 1. PMID 34217637